CLINICAL TRIAL: NCT04495738
Title: Infant Formula and Toddler Drink Feeding Intervention Through 24 Months of Age
Brief Title: Infant Formula and Toddler Drink Feeding Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in research focus
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AL38
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Respiratory Infections in Children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Feeding Group (Active Comparator): Ready to feed milk-based product
  Interventions: Other: Control Infant Formula; Other: Control Toddler Drink
- Experimental Feeding Group (Experimental): Ready to feed milk-based product with oligosaccharides
  Interventions: Other: Experimental Infant Formula; Other: Experimental Toddler Drink
- Human Milk (HM) Reference Group (Other): HM from infant's own mother and as needed supplemental infant formula and toddler milk-based product
  Interventions: Other: Supplemental Formula for HM Group; Other: Toddler Drink for HM group

INTERVENTIONS:
Other: Control Infant Formula — Ad libitum or as instructed by HCP, feeding period from enrollment to 12 months of age
  Arms: Control Feeding Group
Other: Control Toddler Drink — 16 fl oz per day as primary milk beverage; feeding period from 12 to 24 months of age
  Arms: Control Feeding Group
Other: Experimental Infant Formula — Ad libitum or as instructed by HCP, feeding period from enrollment to 12 months of age
  Arms: Experimental Feeding Group
Other: Experimental Toddler Drink — 16 fl oz per day as primary milk beverage; feeding period from 12 to 24 months of age
  Arms: Experimental Feeding Group
Other: Supplemental Formula for HM Group — Ad libitum formula given up to 12 months of age if HM is supplemented
  Arms: Human Milk (HM) Reference Group
Other: Toddler Drink for HM group — 16 fl oz per day if weaned from HM feedings
  Arms: Human Milk (HM) Reference Group

SUMMARY:
The purpose of this randomized, multi-center, controlled, double-blind, parallel study is to evaluate the health and developmental outcomes of children fed a new infant formula and toddler drink through 24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Participant is judged to be in good health as determined from participant's medical history
* Participant is a singleton from a full-term birth with a gestational age of 37 - 42 weeks
* Participant's birth weight was ≥ 2490 g (~5 lbs. 8 oz.)
* If parent(s) elect to formula feed the participant they confirm their intention to feed their participant the study product as the sole source of feeding until 4 months of age, and as the sole milk beverage during the first 12 months of life
* If parent(s) elect to formula feed the participant, they confirm their intention to feed the participant the assigned toddler drink from 12 months of life to 24 months of life as the primary milk beverage
* If parent(s) elect to feed the participant mother's human milk, they confirm that their infant was exclusively fed mother's human milk since birth and confirm their intention to continue exclusively feeding human milk as the sole source of feeding through 4 months of age
* If parent(s) of human milk fed participant elect to supplement or wean after 4 months to 24 months of age, they confirm their intention to use the supplemental/weaning formula or toddler drink as the primary milk beverage
* Parent(s) of formula-fed participant confirm their intention not to administer vitamin or mineral supplements, from enrollment through the duration of the study
* Parent(s) confirm their intention not to administer solid foods or juices to the participant from enrollment through 6 months of age
* Participant's parent(s) has voluntarily signed and dated an informed consent form (ICF), approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC) and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study.

Exclusion Criteria:

* An adverse maternal, fetal or participant medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development
* Participant is taking and plans to continue medications (including over the counter (OTC), home remedies, herbal preparations, prebiotics or probiotics, or rehydration fluids that might affect GI tolerance
* Participant is in another study that has not been approved as a concomitant study
* Participant has been treated with antibiotics prior to enrollment

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Incidence of respiratory infection between study groups | Study Day 1 to 6 Months of Age
  Adverse event reports

SECONDARY OUTCOMES:
Infection morbidity between study groups | Study Day 1 to 24 Months of Age
  Adverse event reports

OTHER OUTCOMES:
Weight | Study Day 1 to 24 Months of Age
  Weight in grams
Length | Study Day 1 to 24 Months of Age
  Length in cm
Head Circumference (HC) | Study Day 1 to 24 Months of Age
  HC in cm
Gastrointestinal Tolerance | Study Day 1 to 119 Days of Age
  Parent completed diary
Dietary Intake | Study Day 1 to 24 Months of Age
  Parent completed diary
Infant Feeding and Stool Patterns Questionnaire | 28 Days of Age to 119 Days of Age
  Parent completed questionnaire; 16, 5-point Likert scale questions, scaled in the negative direction
Infant Behavior Questionnaire | 119 Days of Age
  Parent completed questionnaire; 22 questions with 5-point Likert scale questions, scaled in the negative direction
Formula Satisfaction Questionnaire | 28 Days of Age to 6 Months of Age
  Parent completed questionnaire; 12 questions with 5-point Likert scale questions scaled in the negative direction
Toddler Drink Satisfaction Questionnaire | 15 Months of Age to 24 Months of Age
  Parent completed questionnaire; 12 questions with 5-point Likert scale questions scaled in the negative direction
Human Milk Sample | 84 Days of Age
  Oligosaccharide characterization
Stool Sample | Study Day 1 to 24 Months of Age
  Microbiota characterization
Saliva Sample | 84 Days of Age
  Maternal-Infant secretor status
Modified Home Short Form | 6 Months of Age to 24 Months of Age
  Parent completed questionnaire; 8 questions related to the home environment adapted from the HSF compared between groups
Behavioral Questionnaire | 12 Months of Age to 24 Months of Age
  Parent completed questionnaire; 8 questions related to sleep, physical activity and screen time
Ages & Stages Questionnaire | 6 Months of Age to 18 Months of Age
  Parent completed questionnaire; 5 Developmental areas; Scores to the six questions in each area are totaled; Higher scores indicate more positive outcomes
Bayley Scale of Infant & Toddler Development | 12 Months of Age to 24 Months of Age
  Examiner rated assessment; Scores are totaled and compared to normative age group data and between groups
MacArthur Communicative Developmental Inventory | 12 Months of Age to 24 Months of Age
  Parent completed questionnaire of Words and Gestures and Words and Sentences; Percentiles compared to normative group data and between groups
Edinburgh Postnatal Depression Scale | 28 Days of Age
  Mother completed questionnaire; Scores for each of the 10 items are totaled; Higher scores indicate more depressive symptoms
Medications | Study Day 1 to 24 Months of Age
  Medication usage including frequency and reason for use
Adverse Events | Study Day 1 to 24 Months of Age
  Standard Adverse Event reporting
Health Resource Utilization | Study Day 1 to 24 Months of Age
  Number of visits

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Barrett Reis, PhD, RD, Study Chair — Abbott Nutrition
Locations (27):
- United States (27):
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Eclipse Clinical Research, Tucson, Arizona
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Boeson Research 3266, Grand Junction, Colorado
  - TOPAZ Clinical Research, Inc., Apopka, Florida
  - ASCLEPES Research Centers, Spring Hill, Florida
  - Meridian Clinical Research 3259, Macon, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - Qualmedica Research 3272, Evansville, Indiana
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Qualmedica Research, LLC 3270, Owensboro, Kentucky
  - Meridian Clinical Research 3080, Baton Rouge, Louisiana
  - Boeson Research 3265, Kalispell, Montana
  - Boeson Research 3267, Missoula, Montana
  - Meridian Clinical Research 3264, Grand Island, Nebraska
  - Meridian Clinical Research 3263, Hastings, Nebraska
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - Holston Medical Group, Kingsport, Tennessee
  - MultiCare Institute for Research & Innovation, Dickinson, Texas
  - Maximos Ob/Gyn, League City, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - PAS Research 3273, McAllen, Texas
  - Multicare Rockwood Pediatrics, Spokane, Washington
  - Mercury Clinical Research 3261, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No